CLINICAL TRIAL: NCT01001403
Title: Effect of Nafamostat Mesilate on Hemodynamic Stability After Reperfusion of the Liver Graft
Brief Title: Effect of Nafamostat on Postreperfusion Syndrome (PRS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Chul Woo Jung, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CWJung_futhan-liver TPL
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Results first posted 2010-05-03 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Liver Transplantation; Postreperfusion Syndrome
MeSH Terms: interventions — nafamostat; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nafamostat (Experimental): The Nafamostat mesilate group received 0.2 mg/kg of nafamostat mesilate intravenously 1 min before reperfusion of the liver graft.
  Interventions: Drug: Nafamostat
- Control (Placebo Comparator): The control group received 10 ml of normal saline (same volume as nafamostat)intravenously 1 min before reperfusion of the liver graft.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Nafamostat — 0.2 mg/kg as bolus 1 minute before reperfusion
  Arms: nafamostat
Drug: Normal saline — 10 ml of normal saline
  Arms: Control

SUMMARY:
This study intends to see the effect of nafamostat on the attenuation of postreperfusion syndrome (PRS) that frequently occurs during liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 year old scheduled to undergo liver transplantation

Exclusion Criteria:

* Previous history of pulmonary, cardiovascular, or renal disease
* Previous history of allergic reactions to nafamostat

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nafamostat | Control
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nafamostat | Control | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 28 | 58
  >=65 years | 1 | 3 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (10) | 52 (11) | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 28 | 25 | 53
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Moderate and Severe Postreperfusion Syndrome (PRS)
Description: Before entering the study, we re-defined the criteria of PRS. From our clinical experiences, two types of PRS were observed according to its severity and treatment option. "Moderate" PRS was identical to previously defined PRS: more than 30% decrease of mean arterial pressure lasting over 1 min was observed within 5 min after reperfusion of the liver graft. However, we differentiated a "severe" form of PRS, in which MAP rapidly fell below 40 mmHg, from the moderate one, because severe PRS required prompt intervention to prevent a permanent damage of vital organs.
Time Frame: during 5 min after reperfusion of liver graft
Measure: Number; unit: participants
Arm/Group | Nafamostat | Control
Number analyzed (Participants) | 31 | 31
participants | 15 | 25

ADVERSE EVENTS:
Arm/Group | Nafamostat | Control
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No